CLINICAL TRIAL: NCT00474656
Title: The Oscillation for ARDS Treated Early (OSCILLATE) Trial Pilot Study
Acronym: OSCILLATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Critical Care Trials Group (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); McMaster University (Other); University of Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 164451
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: high frequency oscillation; lung-protective ventilation; ARDS; ventilator-induced lung injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury | interventions — High-Frequency Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: High-frequency oscillation
Device: Conventional lung-open mechanical ventilation

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a common and catastrophic complication of critical illness related to burns, motor vehicle accidents, or overwhelming infection. ARDS kills 40-70% of affected patients. Patients with ARDS require life support in the form of a ventilator to breathe for them while their lungs heal. Ironically, ventilators can cause further damage to the lungs. We are conducting a study comparing 2 methods to protect the lungs from further damage. One method uses standard mechanical ventilators and the other uses a new type of ventilator, called a high frequency oscillator. We propose to test whether this high frequency oscillation will reduce the relative risk of dying from ARDS. 72 patients from 12 intensive care units in Canada and Saudi Arabia will participate in this preliminary study to test the feasibility of our study methods. If feasible, we plan to move on and conduct a large multinational study to definitively answer this question.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex, 16 years and above;
* Acute onset of respiratory failure, with fewer than 2 weeks of new pulmonary symptoms;
* Endotracheal intubation or tracheostomy;
* Hypoxaemia - defined as a PaO2/FiO2 ≤ 200 mm Hg;
* Bilateral alveolar consolidation (airspace disease) seen on frontal chest radiograph

Exclusion Criteria:

* Remaining duration of mechanical ventilation < 48 hours, as judged by the attending physician;
* Primary cause of acute respiratory failure judged by attending physician to be cardiac in origin;
* Lack of commitment to ongoing life support;
* Weight < 35 kg;
* Severe chronic respiratory disease
* Morbid obesity - defined as > 1 kg / cm body height;
* Neurological conditions with risk of intracranial hypertension (hypercapnia should be avoided);
* Neuromuscular disease that will result in prolonged need for mechanical ventilation;
* Previous enrolment in this trial;
* All inclusion criteria present for > 72 hours;
* On HFO at the time of screening.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-06; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
adherence to our explicit mechanical ventilation protocols; | duration of mechanical ventilation
to measure and understand the reasons for crossovers between groups | duration of mechanical ventilation
to estimate the rate of patient recruitment, and understand barriers to recruitment
to document our ability to achieve close to complete follow-up for mortality and quality of life in the 6 months following enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Niall D Ferguson, MD, MSc, Principal Investigator — University of Toronto; Maureen O Meade, MD, MSc, Principal Investigator — McMaster University
Locations (12):
- Canada (11):
  - University of Alberta Medical Centre, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - St Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Mt Sinai Hospital, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
- King Fahad National Guard Hospital, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Arabi YM, Cook DJ, Zhou Q, Smith O, Hand L, Turgeon AF, Matte A, Mehta S, Graham R, Brierley K, Adhikari NK, Meade MO, Ferguson ND; Canadian Critical Care Trials Group. Characteristics and Outcomes of Eligible Nonenrolled Patients in a Mechanical Ventilation Trial of Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2015 Dec 1;192(11):1306-13. doi: 10.1164/rccm.201501-0172OC. PMID 26192398
- [Derived] Ferguson ND, Cook DJ, Guyatt GH, Mehta S, Hand L, Austin P, Zhou Q, Matte A, Walter SD, Lamontagne F, Granton JT, Arabi YM, Arroliga AC, Stewart TE, Slutsky AS, Meade MO; OSCILLATE Trial Investigators; Canadian Critical Care Trials Group. High-frequency oscillation in early acute respiratory distress syndrome. N Engl J Med. 2013 Feb 28;368(9):795-805. doi: 10.1056/NEJMoa1215554. Epub 2013 Jan 22. PMID 23339639